CLINICAL TRIAL: NCT03546309
Title: Safety and Efficacy of Remote Ischemic Conditioning in Pediatric Moyamoya Disease Patients Treated With Revascularization Therapy
Brief Title: Safety and Efficacy of RIC in Pediatric Moyamoya Disease Patients Treated With Revascularization Therapy
Acronym: RIC-PMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: The Fifth Medical Center of the Chinese People's Liberation Army (PLA) General Hospital (Unknown)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIC-PMD
Record Dates: First submitted 2018-03-12; First posted 2018-06-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Moyamoya Disease; Pediatric
Keywords: pediatric moyamoya disease; remote ischemic conditioning; revascularization therapy
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): Patients allocated to the RIC group will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 50 mmHg over systolic blood pressure for five cycles of 5 min followed by 5 min of relaxation of the cuffs.They will also accept medication treatment by professional neurologists.
  Interventions: Device: RIC group
- Medication group (Other): Patients allocated to the medication group will accept medication treatment by professional neurologists.
  Interventions: Other: Medication group

INTERVENTIONS:
Device: RIC group — Patients allocated to the RIC group will undergo RIC procedure during which bilateral arm cuffs are inflated to a pressure of 50 mmHg over systolic blood pressure for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Arms: RIC group
Other: Medication group — Patients allocated to Medication group will accept medication treatment by professional neurologists
  Arms: Medication group

SUMMARY:
Revascularization surgery has been the standard treatment to prevent ischemic stroke in pediatric Moyamoya disease (MMD) patients with ischemic symptoms. However, perioperative complications, such as hyperperfusion syndrome, new infarct on imaging, or ischemic stroke, are inevitable. Remote ischemic conditioning (RIC) is a noninvasive and easy-to-use neuroprotective strategy, and it has potential effects on preventing hyperperfusion syndrome and ischemic infarction.

DETAILED DESCRIPTION:
This study will provide insights into the preliminary proof of principle, safety, and efficacy of RIC in pediatric MMD patients undergoing revascularization surgery therapy, and this data will provide parameters for future larger scale clinical trials if efficacious.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥0 and ≤18
* All of the patients underwent digital subtraction angiography and met the current diagnostic criteria recommended by the Research Committee on MMD (Spontaneous Occlusion of the Circle of Willis) of the Ministry of Health and Welfare of Japan in 2012
* Suzuki stages concentrated in Stage III and IV
* Presentation with ischemic symptoms, such as transient ischemic attack (TIA), headache, seizure, hemorrhagic stroke, and ischemic stroke confirmed by MRI
* Informed consent obtained from patient or acceptable patient's surrogate

Exclusion Criteria:

* Severe hepatic or renal dysfunction
* Severe hemostatic disorder or severe coagulation dysfunction
* Patients with unilateral MMD or the presence of secondary moyamoya phenomenon caused by autoimmune disease, Down syndrome, neurofibromatosis, leptospiral infection, or previous skull-base radiation therapy
* Any of the following cardiac disease - rheumatic mitral and or aortic stenosis, prosthetic heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, patent foramen ovale, left ventricular mural thrombus or valvular vegetation, congestive heart failure, bacterial endocarditis, or any other cardiovascular condition interfering with participation
* Serious, advanced, or terminal illnesses with anticipated life expectancy of less than one year
* Patient participating in a study involving other drug or device trial study
* Patients with existing neurological or psychiatric disease that would confound the neurological or functional evaluations
* Unlikely to be available for follow-up for 3 months
* Contraindication for RIC - severe soft-tissue injury, fracture, or peripheral vascular disease in the upper limbs.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
the incidence of major neurologic complications | during the perioperative period
  Including transient ischemic attack, cerebral infarction, intracranial hemorrhage, and seizures.

SECONDARY OUTCOMES:
The score of National Institute of Health stroke scale score | change from baseline (preoperation) at 24 hours, 48 hours, 72 hours, and at 5-7 days or if discharged earlier
  National Institute of Health Stroke Scale (NIHSS) is considered as a standardized assessment of neurological functions in the acute phase of stroke, and it is generally used to quantify patient's neurological impairments on 15 items in 11 fields of different neurological status.The score of the scale ranges from 0 to 42.And higher score indicates worse neurological function.
The score of Modified Rankin scale score | change from baseline (pre-RIC treatment) at 180 days after revascularization therapy
  The Modified Rankin Scale Score (mRS) is the most comprehensive and most widely used primary outcome measurement to assess the neurological functional disability in contemporary acute stroke trials. The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranges from 0 (no symptom) to 5 (severe disability) and 6 (death). We will use mRS to evaluate the degree of disability or dependence during daily activities. The mRS will be assessed by certified study investigator, who is blinded to the treatment assignment, at 90 days postoperation. The distribution of mRS will be compared between groups
Symptomatic intracerebral hemorrhage | during the first 180 days after revascularization therapy
  Symptomatic intracranial hemorrhage, including any subarachnoid hemorrhage associated with clinical symptoms and symptomatic intracerebral hemorrhage. Head computed tomography or magnetic reasoning imaging (MRI) scan will be performed to confirm intracerebral hemorrhage, and the imaging will be evaluated by two independent neuroradiologists who are blinded to the study assignment.
Incidence of new infarct in brain | during 72 hours and 180 days after revascularization therapy
  Head MRI is a precise method which is commonly used to evaluate weather there's new infarct in brain.
Angiographic outcome | 180 days after revascularization therapy
  Angiographic outcome will be assessed following Matsushima's criteria (proportion of the middle cerebral artery territory with revascularization from collaterals from the external carotid artery through the burr holes): Grade A: >2/3; Grade B: between 1/3 and 2/3; Grade C: <1/3.
Death and adverse event | 180 days after revascularization therapy
  All causes of death will be included to compute mortality at 180 days postoperation, and mortality will be compared between groups. Any adverse event will be reported and its relationship with the RIC intervention will be evaluated.
Infarct volume in brain | during 72 hours and 180 days after revascularization therapy
  Head MRI is a precise method which is commonly used to evaluate infarct size.
Distal radial pulses | within 7 days after RIC treatment
  professional doctors will check the distal radial pulses
Visual inspection for local edema | within 7days after RIC treatment
  Professional oculists will check the fundus oculi to evaluate whether there is local edema.
The number of patients with erythema,and/or skin lesions related to RIC | within 7days after RIC treatment
  Professional doctors will check it and the investigator will record the number.
Palpation for tenderness | within 7days after RIC treatment
  Professional doctors will check it.
The number of patients not tolerating RIC procedure,and refuse to continue the RIC procedure | within 7days after RIC treatment
  The investigator will record the number.
The number of patients with any other adverse events related to RIC intervention | within 7days after RIC treatment
  The investigator will record the number.
The score of ABCD2 | change from baseline (pre-RIC treatment) at 180 days after revascularization therapy
  We use this scale to evaluate the patients' risk of stroke who with TIA .The score of the scale ranges from 0 to 7, and the higher score indicates higher risk of stroke in the patients who with TIA.The scale will be assessed by qualified investigator who are blinded to the treatment assignment
The level of S-100A4 | change from baseline (pre-RIC treatment) at 7 days after RIC treatment, 24 (-6/+12) hours, 72 ± 6 hours and 6 months postoperation
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of matrix metalloproteinase 9 (MMP-9) | change from baseline (pre-RIC treatment) at 7 days after RIC treatment, 24 (-6/+12) hours, 72 ± 6 hours and 6 months post-operation
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of basic fibroblast growth factor | change from baseline (pre-RIC treatment) at 7 days after RIC treatment, 24 (-6/+12) hours, 72 ± 6 hours and 6 months post-operation
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of platelet derived growth factor | change from baseline (pre-RIC treatment) at 7 days after RIC treatment, 24 (-6/+12) hours, 72 ± 6 hours and 6 months post-operation
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
The level of vascular endothelial growth factor | change from baseline (pre-RIC treatment) at 7 days after RIC treatment, 24 (-6/+12) hours, 72 ± 6 hours and 6 months post-operation
  Blood samples will be drawn from cubital vein to test these biomarkersThese samples will be centrifuged immediately after collection and stored at - 80 until batch evaluation
the score of PSQI | 0-30 days
  The Pittsburgh Sleep Quality Index (PSQI) is a standardized questionnaire used to assess sleep quality and disturbances over a one-month time interval.
the score of SNAP-IV | 0-30 days
  SNAP-IV (Swanson, Nolan, and Pelham Teacher and Parent Rating Scale) is a widely used assessment tool designed to evaluate behavioral and emotional problems in children and adolescents.
cerebral perfusion status | 0-3 months
  cerebral perfusion status in the operation side at 3 months posttreatment as assessed by magnetic resonance perfusion

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuriyama S, Kusaka Y, Fujimura M, Wakai K, Tamakoshi A, Hashimoto S, Tsuji I, Inaba Y, Yoshimoto T. Prevalence and clinicoepidemiological features of moyamoya disease in Japan: findings from a nationwide epidemiological survey. Stroke. 2008 Jan;39(1):42-7. doi: 10.1161/STROKEAHA.107.490714. Epub 2007 Nov 29. PMID 18048855
- [Background] Kim SK, Seol HJ, Cho BK, Hwang YS, Lee DS, Wang KC. Moyamoya disease among young patients: its aggressive clinical course and the role of active surgical treatment. Neurosurgery. 2004 Apr;54(4):840-4; discussion 844-6. doi: 10.1227/01.neu.0000114140.41509.14. PMID 15046649
- [Background] Kim JE, Oh CW, Kwon OK, Park SQ, Kim SE, Kim YK. Transient hyperperfusion after superficial temporal artery/middle cerebral artery bypass surgery as a possible cause of postoperative transient neurological deterioration. Cerebrovasc Dis. 2008;25(6):580-6. doi: 10.1159/000132205. Epub 2008 May 16. PMID 18483458
- [Background] Fujimura M, Shimizu H, Inoue T, Mugikura S, Saito A, Tominaga T. Significance of focal cerebral hyperperfusion as a cause of transient neurologic deterioration after extracranial-intracranial bypass for moyamoya disease: comparative study with non-moyamoya patients using N-isopropyl-p-[(123)I]iodoamphetamine single-photon emission computed tomography. Neurosurgery. 2011 Apr;68(4):957-64; discussion 964-5. doi: 10.1227/NEU.0b013e318208f1da. PMID 21221039
- [Background] Funaki T, Takahashi JC, Takagi Y, Kikuchi T, Yoshida K, Mitsuhara T, Kataoka H, Okada T, Fushimi Y, Miyamoto S. Unstable moyamoya disease: clinical features and impact on perioperative ischemic complications. J Neurosurg. 2015 Feb;122(2):400-7. doi: 10.3171/2014.10.JNS14231. Epub 2014 Nov 28. PMID 25423271
- [Background] Zhao W, Meng R, Ma C, Hou B, Jiao L, Zhu F, Wu W, Shi J, Duan Y, Zhang R, Zhang J, Sun Y, Zhang H, Ling F, Wang Y, Feng W, Ding Y, Ovbiagele B, Ji X. Safety and Efficacy of Remote Ischemic Preconditioning in Patients With Severe Carotid Artery Stenosis Before Carotid Artery Stenting: A Proof-of-Concept, Randomized Controlled Trial. Circulation. 2017 Apr 4;135(14):1325-1335. doi: 10.1161/CIRCULATIONAHA.116.024807. Epub 2017 Feb 7. PMID 28174194